CLINICAL TRIAL: NCT04119284
Title: Safety and Efficacy of a Vertebral Body Tethering Technique for Pediatric Idiopathic Scoliosis
Brief Title: Safety Outcomes of Vertebral Body Tethering Technique
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB suspended the study.
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Suken Shah, PI, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1365311; G180238 (Other: FDA)
Record Dates: First submitted 2019-09-27; First posted 2019-10-08 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Adolescent Scoliosis
Keywords: scoliosis; Vertebral Body Tethering; curve; Shah
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Anterior Vertebral Tethering (Experimental): Anterior Vertebral Tether Vertebral body tethering done through anterior spine surgery under anesthesia.
  Interventions: Device: Anterior body tether (ABT)

INTERVENTIONS:
Device: Anterior body tether (ABT) — To insert the ABT in patients to correct AIS.
  Other Names: Reflect/Transition™ Stabilization System Polyethylene terephthalate (PET) cord

SUMMARY:
The objectives of this study is to assess whether the intervention (Anterior Vertebral Tethering) is a safe and efficacious method of anterior approach surgery for spinal deformity in pediatric scoliosis.

DETAILED DESCRIPTION:
Scoliosis is a condition where the spine is deformed by a curvature in the coronal plane. It is generally associated with a twisting (axial plane) deformity as well.

Curves between 10 and 25 degrees are considered mild. Curves between 25- and 50 degrees are classified as moderate. Curves greater than 50 degrees are termed severe. The current standard of care for moderate Adolescent Idiopathic Scoliosis(AIS) in patients with remaining growth is to utilize a thoracolumbosacral orthosis (TLSO brace) to prevent progression of deformity. The scientific evidence has supported the efficacy of this intervention in avoiding progression of the Cobb angle to 50 degrees or more.

If treated with a TLSO brace, many idiopathic scoliosis patients would conceivably be subjected to years of brace wear and the cost and psychological factors inherent therein. Additional downsides of brace treatment include the potentially negative psychosocial impact of wearing an external sign of deformity during adolescence, a key period of emotional development. Prior research has identified negative psychosocial effects related to wearing a brace in children.

Recent evidence has suggested that certain curve patterns will likely progress to 50 degrees or more, despite treatment with a TLSO brace. Sanders, et al. demonstrated a correlation of Cobb angle (greater than 35 degrees) and skeletal maturity (bone age 4 or less) to the risk of progression to 50 degrees or more, despite TLSO bracing. The evidence supports that the current practice of TLSO bracing is not an effective treatment to avoid progression to 50 degrees in these patients. It is on this population (thoracic Cobb angle greater than 35 degrees, bone age of 4 or less) that we intend to test the safety and efficacy of Anterior Vertebral Body Tethering to avoid curve progression to more than 50 degrees.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 8 to 16 years old at time of enrollment (inclusive)
2. Diagnosis of idiopathic scoliosis
3. Sanders bone age of less than or equal to 4
4. Thoracic curve of greater than or equal to 35 degrees and less than or equal to 60 degrees
5. Lumbar curve less than 35 degrees
6. Patient has already been identified for and recommended to have surgical intervention
7. Spina bifida occulta is permitted
8. Spondylolysis or Spondylolisthesis is permitted, as long as it is non-operative, the subject has not had any previous surgery for this, and no surgery is planned in the future

Exclusion Criteria:

1. Pregnancy (current)
2. Prior spinal or chest surgery
3. MRI abnormalities (including syrinx greater than 4mm, Chiari malformation, or tethered cord)
4. Neuromuscular, thoracogenic, cardiogenic scoliosis, or any other non-idiopathic scoliosis
5. Associated syndrome, including Marfan syndrome or neurofibromatosis
6. Sanders bone age greater than 4
7. Thoracic curve less than 35 degrees or greater than 60 degrees
8. Lumbar curve greater than or equal to 35 degrees
9. Unable or unwilling to firmly commit to returning for required follow-up visits
10. Investigator judgement that the subject/family may not be a candidate for the intervention

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suken Shah, MD, Principal Investigator — Nemours-AIDHC
Locations (1):
- Nemours Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Informed Consent Form — http://irbnet.org — The Informed consent form can be obtained while the patient is seen for scoliosis at Nemours-AIDHC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anterior Vertebral Tethering
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anterior Vertebral Tethering
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 11.34 [9.33 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Cobb angle [Mean (Full Range); unit: degree] — Cobb angle is measured in degrees on x-rays.
  degree | 48.125 [42 to 55]

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events After the Procedure
Description: We will look for any changes in neurological status, tether failure, implant reoperation, overcorrection and wound infections.
  Adverse events will be summarized by their severity and frequency and reported to IRB and Data Safety board on timely bases.
  The PI will determine if these events are related to the device.
Time Frame: 2 years after the surgery
Measure: Number; unit: Number of Tether failures
Arm/Group | Anterior Vertebral Tethering
Number analyzed (Participants) | 8
Number of Tether failures | 8

2. Secondary Outcome: Cobb Angle in Degrees
Description: The difference between pre and post-operative Cobb angle measurements.
Time Frame: The difference between Cobb angles measured prior to surgery and 2 years past surgery.
Population: 8 patients completed the study. Their pre-operative main curve measurements (Cobb angles) were measured and summarized. The same measurements were obtained at the 2 years follow up visits. The data was summarized and the means difference with the standard deviation were reported.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anterior Vertebral Tethering
Number analyzed (Participants) | 8
degrees | 22.37 (4.16)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Anterior Vertebral Tethering
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anterior Vertebral Tethering (N=8)
Broken Tether (Surgical and medical procedures) | 8 (8) — The tether device broke or suspectedly broke past one year out of surgery based on x-ray images.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT04119284/Prot_SAP_001.pdf